CLINICAL TRIAL: NCT02781662
Title: Improving Safety After Hospitalization in Older Persons on High-Risk Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Reliant Medical Group (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R18HS023774 (AHRQ); R18HS023774 (AHRQ)
Record Dates: First submitted 2016-05-09; First posted 2016-05-24 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Medication Safety
Keywords: Safety; Hospitalization; Older Persons; High-Risk

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No Intervention; Control Arm: Receives Written Medication Information
- Intervention (Experimental): Behavioral: Pharmacist Home-Visit
  Interventions: Behavioral: Pharmacist Home-Visit

INTERVENTIONS:
Behavioral: Pharmacist Home-Visit
  Arms: Intervention

SUMMARY:
This study evaluates an intervention to reduce medication errors and adverse drug events in older adults who have recently been discharged from the hospital and prescribed anticoagulants, diabetes agents, or opioids. Half of the study participants will receive the intervention, while the other half will receive usual care.

DETAILED DESCRIPTION:
The overarching objective of this research study is to pursue a large randomized controlled trial (RCT) focused on older patients recently discharged from the hospital who have been prescribed medications within one of three high-priority, high-risk drug classes in order to reduce the risk of clinically important medication errors. The National Action Plan for Adverse Drug Event (ADE) Prevention identified three high-priority drug classes as key targets for reducing the risk of drug-related injuries: anticoagulants; diabetes agents (insulin and oral agents); and opioids. These medication classes were chosen because they account for the greatest number of measurable drug-related harms to patients, and a substantial proportion of ADEs associated with these medications is considered preventable. The clinical trial will determine the value of a multifaceted medication error and ADE reduction intervention with a special focus on in-home assessment.

Components of the intervention will include: (1) in-home assessment of high-risk patients by a clinical pharmacist; (2) best-practice, evidence-based medication safety tools and resources targeted to high-risk patients and their caregivers; (3) communication with the primary care team via the electronic health record (EHR) regarding concerns relevant to the use of high-risk medications as well as other medication safety concerns; and (4) a follow-up phone call by the pharmacist to the patient and/or caregiver within 14 days of the home visit. The primary outcome of interest will be clinically important medication errors, a composite outcome comprised of preventable or ameliorable ADEs and potential ADEs due to medication discrepancies or non-adherence. Secondary outcomes will include: (1) preventable or ameliorable ADEs; (2) potential ADEs due to discrepancies or non-adherence; and (3) preventable or ameliorable ADEs judged to be serious, life-threatening, or fatal.

The specific aims for our study are as follows:

Aim 1: To adapt and integrate existing "best-practice," evidence-based medication safety tools, resources, and approaches into a cohesive, multifaceted intervention to reduce the occurrence of clinically important medication errors in older adults recently discharged from the hospital using one or more of the three high-priority, high-risk drug classes (anticoagulants, diabetes agents, and opioids).

Aim 2: To assess the impact of the multifaceted intervention on the incidence of clinically important medication errors employing a randomized controlled trial (RCT) design.

Aim 3: To conduct a process evaluation assessing intervention fidelity, adaptation, mechanisms of impact, essential components, and the influence of contextual factors.

Aim 4: To create: 1) a plan for disseminating study findings to stakeholders who might implement the intervention or make decisions about its future use; and 2) an implementation toolkit for those who wish to implement the intervention in practice.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age and having been prescribed one of the three high-risk drug categories (anticoagulants, diabetes agents, and opioids) at the time of hospital discharge and must meet one or more of following screening Items:

  * Prescribed >2 high-risk medications
  * Low health literacy
  * Caregiver (an affirmative response to "Have you received assistance from one or more caregivers over the past 4 weeks?").
  * Low adherence
  * Using >7 different medications

Exclusion Criteria:

* Plans to enroll in hospice upon discharge.
* Discharged for a psychiatric condition.
* Discharged to a skilled nursing facility, rehabilitation hospital, or nursing home.
* Patient is not capable of providing informed consent, and a proxy is not available.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Clinically important medication errors (preventable drug events and potential adverse events due to medication discrepancies or non-adherence). | Within 45 days subsequent to hospital discharge
  To assess for the occurrence of clinically important medication errors, the investigators will use methods that they have developed, tested, and validated in previous investigations relating to drug-related incidents. Two pharmacist-investigators, who will not be involved in the intervention, will screen for signals of possible clinically important medication errors in the patient's electronic health record and in a structured telephone interview. The semi-structured telephone interview will be conducted according to the approach used by Forester, et. al (Forster AJ, Murff HJ, Peterson JF, et al. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003; 138(3):161-167).

CONTACTS AND LOCATIONS:
Overall Officials: Jerry H Gurwitz, MD, Principal Investigator — Meyers Primary Care Institute, University of Massachusetts Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gurwitz JH, Kapoor A, Garber L, Mazor KM, Wagner J, Cutrona SL, Singh S, Kanaan AO, Donovan JL, Crawford S, Anzuoni K, Konola TJ, Zhou Y, Field TS. Effect of a Multifaceted Clinical Pharmacist Intervention on Medication Safety After Hospitalization in Persons Prescribed High-risk Medications: A Randomized Clinical Trial. JAMA Intern Med. 2021 May 1;181(5):610-618. doi: 10.1001/jamainternmed.2020.9285. PMID 33646267